CLINICAL TRIAL: NCT07332468
Title: Digital Remote Management for Care and Continuous Optimization Versus Usual Care to Reduce Risk of Atherosclerotic Cardiovascular Diseases (DigiCare-ASCVD)
Acronym: DigiCare-ASCVD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of cardiology department, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2025288
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerotic Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care Group (No Intervention): Usual Care Group: Patients receive standard BP, lipids,glucose and physical activity management including guideline-directed medication and outpatient follow-up at 3, 6, 9, 12 months.
- Digital Remote Management Group (Experimental): In addition to usual care, patients receive a 1-year intervention via a smartphone-based ""physician-machine collaboration"" platform：
  1. BP Management: Daily or weekly self-monitoring based on control status. System triggers alerts for BP >130/80 mmHg and generates medication adjustment suggestions for physician approval.
  2. Lipid Management: Reminder for lab tests. OCR technology parses results. If LDL-C ≥2.6 mmol/L, the system suggests regimen intensification for physician review.
  3. Blood Glucose Management: Reminder for lab tests. OCR technology parses results.If Fasting Blood Glucose (FBG) ≥6.1 mmol/L for patients without diabetes and FBG ≥7.0 mmol/L for patients with diabetes, the system suggests regimen intensification for physician review.
  4. Medication Management: Daily app-based reminders and clock-in tasks. Non-adherence triggers automated reminders and human follow-up.
  5. Health Education: Regular push of targeted articles/videos on secondary prevention。
  Interventions: Other: Digital Remote Management Group

INTERVENTIONS:
Other: Digital Remote Management Group — In addition to usual care, patients receive a 1-year intervention via a smartphone-based ""physician-machine collaboration"" platform：
  1. BP Management: Daily or weekly self-monitoring based on control status. System triggers alerts for BP >130/80 mmHg and generates medication adjustment suggestions for physician approval.
  2. Lipid Management: Reminder for lab tests. OCR technology parses results. If LDL-C ≥2.6 mmol/L, the system suggests regimen intensification for physician review.
  3. Blood Glucose Management: Reminder for lab tests. OCR technology parses results.If Fasting Blood Glucose (FBG) ≥6.1 mmol/L for patients without diabetes and FBG ≥7.0 mmol/L for patients with diabetes, the system suggests regimen intensification for physician review.
  4. Medication Management: Daily app-based reminders and clock-in tasks. Non-adherence triggers automated reminders and human follow-up.
  5. Health Education: Regular push of targeted articles/videos on secondary prevention。
  Arms: Digital Remote Management Group

SUMMARY:
The DigiCare-ASCVD study is an investigator-initiated, multicenter, open-label, parallel-group randomized controlled trial. It aims to evaluated whether digital remote management is superior to usual care in reducing risk of atherosclerotic cardiovascular diseases and improving blood pressure control, glycemic control, lipids control, medication compliance and lifestyle.

DETAILED DESCRIPTION:
"Atherosclerotic cardiovascular disease (ASCVD) is a leading global cause of mortality. Primary care is central to its prevention within tiered healthcare systems, yet faces challenges including physician training gaps and inefficient specialist referrals. Digital remote interventions offer a promising solution due to widespread smartphone/internet access, enabling convenient care and real-time data use. Current tools focus on patient education/reminders or clinical decision support (CDSS) separately. However, effective long-term ASCVD management requires an integrated system that combines CDSS-guided treatment with comprehensive, sustained risk-factor monitoring (e.g., blood pressure, lipids). This study aims to develop and validate such an integrated remote management platform to overcome multi-level barriers, disseminate advanced resources to primary care, and enhance equitable cardiovascular risk prevention.

The DigiCare-ASCVD Study is a multicenter, open-label, randomized controlled trial with a 1:1 parallel-group design. It will enroll 790 patients at high risk for ASCVD. All enrolled patients will be randomly assigned in a 1:1 ratio to either the Digital Remote Management group or the usual care group.

Patients in the Digital Remote Management group will utilize a smartphone-based ""physician-machine collaboration"" platform. This system integrates home monitoring to track BP, lipids,glucose, medication compliance and physical activity. It features AI-driven alerts for abnormal values, automated medication adjustment suggestions (verified by physicians), and targeted health education The primary endpoint is the mean change in the patient's 10-year ASCVD risk, calculated using the China-PAR risk prediction model, from baseline to the 12-month follow-up."

ELIGIBILITY:
Inclusion Criteria:

1. 10-year ASCVD risk ≥ 10%, calculated using the China-PAR risk prediction model
2. Adultd aged ≥ 35 years
3. Able to use a smartphone (or assisted by family) and agrees to remote management
4. Signed informed consent

Exclusion Criteria:

1. History of acute myocardial infarction, stroke, heart failure, malignant arrhythmia, or prior percutaneous coronary intervention or coronary artery bypass grafting surgery
2. Moderate to severe hepatic dysfunction (Child-Pugh class B-C)
3. CKD stages 4-5 (eGFR <30 ml/min/1.73m²) or on dialysis
4. Chronic obstructive pulmonary disease requiring ongoing home oxygen therapy or chronic oral steroid therapy as an outpatient
5. Pregnant, planning to become pregnant within the next 12 months
6. Life expectancy <12 months (e.g., advanced malignancy, etc.);
7. Cognitive impairment or communication disorder.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in the patient's 10-year ASCVD risk, calculated using the China-PAR risk prediction model | 12 Months

SECONDARY OUTCOMES:
Mean change in the patient's lifetime ASCVD risk, calculated using the China-PAR risk prediction model. | Baseline and 12 Months
Simultaneous Control Rate of Blood Pressure | 12 Months
  SBP < 130 mmHg, DBP < 80 mmHg
Mean change in SBP and DBP compared to baseline | 12 Months
Overweight or Obesity Rate | 12 Months
Smoking Cessation Rate | 12 Months
  Self-reported complete abstinence from smoking among baseline smokers
Medication Adherence | 12 Months
  MARS-10 scale

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, China, Beijing
  - The First Hospital of Jilin University, Changchun, China, Changchun
  - The First Affiliated Hospital of Dalian Medical University, Dalian, China, Dalian
  - The Second Affiliated Hospital of Nanchang University, Nanchang, China, Nanchang
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China, Shanghai

IPD SHARING:
Plan to Share IPD: No